CLINICAL TRIAL: NCT05724407
Title: Evaluation of the Use of a Diagnostic Assistance Tool of Prognostic and Predictive Marker Scoring System in Breast Cancer
Brief Title: Molecular Signature for Breast Cancer
Acronym: MoSi4BCa
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211593
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard of care: Female patient diagnosed for breast cancer
  Interventions: Other: Diagnostic assistance tool

INTERVENTIONS:
Other: Diagnostic assistance tool — Diagnostic assistance tool for analysis of 5 prognostic and predictive markers of breast cancer (HER2, Ki67 Index, Mitoses, Estrogen Hormone Receptor, Hormone Progesteron receptors hormone of Progesteronereceptor).
  Each anatomo-histopathological slide will be re-read 3 times:
  * Reading 1: first reading by a pathologist in the care setting
    * Reading via the standard care procedure (microscope and physical slides)
  * Reading 2: Second reading by another pathologist from the same center, as part of the research.
    * Reading via the standard procedure of care (microscope and physical slides)
  * Reading 3: Third reading by the initial physician, with the algorithmic tool MoSi4BCa after digitization of the slides by a laboratory technician and after a wash-out period of 2 months.

SUMMARY:
The main objective of this study is to evaluate and compare the diagnostic performance of a diagnostic assistance tool for analysis of 5 prognostic and predictive markers of breast cancer (HER2, Ki67 Index, Mitoses, Estrogen Hormone Receptor, Hormone Progesteron receptors hormone of Progesteronereceptor) integrating an automatic analysis algorithm compared to a reference (gold standard defined as the rereading by at least two different anatomopathologists according to the standard method of care) in order to show the non-inferiority of the automatic analysis algorithm compared to this gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Understanding French
* With symptoms of breast cancer that required a biopsy (microbiopsy or macrobiopsy or surgical biopsy) and pathological examination diagnosing breast cancer
* First diagnosis of invasive breast cancercarcinoma
* Affiliated to a social security system
* Agreeing to participate in the study

Exclusion Criteria:

* Refusal to participate in the study
* Not affiliated to the social security system
* Minor or under legal protection
* Patient with a history of breast cancer
* Patient previously treated for breast cancer
* Patient who has relapsed from breast cancer treatment
* Non ductal or non lobular invasive breast cancer carcinoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female breast cancer patient
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performances | at inclusion
  The diagnostic performance of the automatic marker scoring support tool will be assessed based on the pathologists' gold standard using sensitivity and specificity

SECONDARY OUTCOMES:
Duration of procedure | at inclusion
  Comparison of medical time spent reading the slide and establishing marker identification between the standard of care method (microscope and pathologist alone) and the automatic marker scoring support tool (MoSi4BCa)
Cognitive savings | at inclusion
  The contribution of the tool in terms of cognitive savings will be evaluated using quantitative survey for the pathologists participating in the study.
General comfort of use | at inclusion
  The contribution of the tool in terms of general comfort of use will be evaluated using quantitative survey for the pathologists participating in the study.
Organizational constraints | at inclusion
  The organizational constraints of the integration of the solution will be evaluated using a specific questionnaire dedicated to the pathologists and laboratory technicians who participated in the implementation and preparation of the installations.
inter-rater agreement | at inclusion
  Agreement between pathologists will be assessed using using Kappa coefficient or intraclass correlation coefficient
Diagnostic performances | at inclusion
  Diagnostic performances will be assessed using positive likelihood ratio, negative likelihood ratio, positive predictive value, negative predictive value, and C-index or Area Under the Curve

IPD SHARING:
Plan to Share IPD: Undecided